CLINICAL TRIAL: NCT03181490
Title: Multi-centers Validation of a Circulating Tumor DNA Assay to Differentiate Benign and Malignant Pulmonary Nodules Via Targeted High-throughput DNA Methylation Sequencing
Brief Title: Circulating Tumor DNA Methylation Test to Differentiate Benign and Malignant Pulmonary Nodules
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: AnchorDx Medical Co., Ltd. (Industry); First Affiliated Hospital, Sun Yat-Sen University (Other); Nanfang Hospital, Southern Medical University (Other); Central South University (Other); Xiangya Hospital of Central South University (Other); West China Hospital (Other); Qilu Hospital of Shandong University (Other); The Second Hospital University of South China (Other); Shenzhen People's Hospital (Other); The Fourth Affiliated Hospital of Harbin Medical University (Other); Peking University Cancer Hospital & Institute (Other); Xuanwu Hospital, Beijing (Other); Anhui Chest Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Principle Investigator, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: CCTC1701
Record Dates: First submitted 2017-06-07; First posted 2017-06-08 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Nodule, Solitary
Keywords: Pulmonary Nodule; Solitary
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Circulating Tumor DNA Methylation Test — Methylation profiling by high-throughput bisulfite DNA sequencing in blood sample to differentiate benign and malignant pulmonary nodules

SUMMARY:
Current state-of-the-art lung cancer early screening utilizes low-dose CT scan to identify lung nodules smaller than 3 cm in diameter. However, it's still a clinical challenge to differentiate between malignant and benign nodules.

In previous studies, the investigators had taken the approach of methylation profiling by high throughput bisulfite DNA sequencing in tissue samples to identify specific methylation signatures. The investigators had learned methylation patterns that differentiate malignant vs. benign lesions from tissue samples by in-depth data mining, and then used pattern matching to classify plasma samples.

In this study, the investigators are going to validate the efficacy of ctDNA methylation test for diagnosing early lung cancer by comparing results of the pre-surgery ctDNA methylation test with the post-surgery pathology.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational cohort study and seeks to enroll 1230 participants with pulmonary nodules 5-30mm in diameter.

The assay analyzes the ctDNA methylation profiles of lung cancer-specific biomarkers non-invasively using whole blood specimens collected before invasive surgery.

The performance characteristics(sensitivity and specificity) of the pre-surgery ctDNA methylation test for detection of early lung cancer is evaluated in comparison to post-surgery pathology.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or above
* single pulmonary nodule found by CT scan.
* the diameter of the pulmonary nodule is between 5mm to 30mm.
* plan to accept pneumonectomy due to the pulmonary nodule.
* without any sign of lymphatic or distant metastasis.
* agree to sign informed consent.

Exclusion Criteria:

* pregnant or lactating women.
* the diameter of the pulmonary nodule is more than 30mm
* there are 2 or more pulmonary nodules in one single patient.
* any sign of lymphatic or distant metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-surgery adult patients with single pulmonary nodule found by CT scan.
Sampling Method: Probability Sample
Enrollment: 1490 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
The diagnostic performance of the blood-based assay for differentiating benign and malignant pulmonary nodules early using circulating tumor DNA (ctDNA) methylation analysis by next-generation sequencing (NGS) | 1 year
  The efficacy of the blood-based ctDNA methylation assay comparing with pathologic diagnosis, the gold standard, including sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV).

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (14):
- China (14):
  - Department of Thoracic Surgery, Beijing Cancer Hospital, Beijing
  - Department of Thoracic Surgery, Xuanwu Hospital, Capital Medical University, Beijing
  - Department of Thoracic Surgery, The Second Xiangya Hospital of Central South University, Changsha
  - Department of Thoracic Surgery, Xiangya Hospital, Central South University, Changsha
  - Department of Thoracic Surgery, West China Hospital of Sichuan University, Chengdu
  - Department of Thoracic Surgery, Nanfang Hospital of Southern Medical University, Guangzhou
  - Department of Thoracic Surgery, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Department of Thoracic Surgery, The First Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - Department of Thoracic Surgery, The Forth Affiliated Hospital of Harbin Medical University, Haerbin
  - Department of Thoracic Surgery, Anhui Chest Hospital, Hefei
  - Department of Thoracic Surgery, The Second Hospital，University of South China, Hengyang
  - Department of Thoracic Surgery, Qilu Hospital of Shandong University, Jinan
  - Department of Thoracic Surgery, Jiangsu Province Hospital, Nanjing
  - Department of Thoracic Surgery, Shenzhen People's Hospital, Shenzhen